CLINICAL TRIAL: NCT05912023
Title: Vaping Associated Perioperative Pulmonary Complications - Anesthetic Implications
Brief Title: Perioperative Vaping Complications
Status: Active, not recruiting | Type: Observational
Sponsor: Navy Medical Center San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: NMRTCSD.2023.0006
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Vaping; Complication of Anesthesia
Keywords: Vaping; Hypoxemia; Bronchospasm; Perioperative; Pneumonitis
MeSH Terms: conditions — Vaping; Hypoxia; Bronchial Spasm; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vaping patients: Includes patients that actively vape that are undergoing general anesthesia
- Non-vaping patients: Includes patients that do not actively vape that are undergoing general anesthesia

SUMMARY:
Prospective observational study evaluating the incidence, and qualifying the types, of perioperative pulmonary complications in patients that vape.

DETAILED DESCRIPTION:
The primary objective of our study is to determine the rate at which patients that vape or use e-cigarettes experience perioperative pulmonary complications during and following general anesthesia. Complications of interest will include postoperative atelectasis with hypoxemia necessitating oxygen therapy, pneumothorax, pneumonia, bronchospasm, bronchospasm requiring bronchodilator therapy, exacerbation of underlying pulmonary disease, pneumonia, ARDS, and acute respiratory failure. Hospital course, including prolonged PACU stay, prolonged hospital admission for inpatients, and rate of ICU admissions, will also be investigated.

A secondary objective will be to further investigate and include the relationship between vaping cessation timeline in the preoperative period and the occurrence of PPCs, which is similarly underreported in the literature. Furthermore, the study will assess how effectively anesthesia providers are screening for vaping or e-cigarette use as part of the preoperative evaluation, given that "it is unclear whether anesthesiologists and surgeons routinely ask patients explicitly about vaping" in the pre-operative setting. This lack of representative screening for vaping further obscures an understanding of the relationship between vaping, vaping cessation, and PPCs.

ELIGIBILITY:
Inclusion Criteria:

* Surgical Patient
* General Anesthesia
* Hx of vaping
* Age ≥12

Exclusion Criteria:

* Age <12
* Pregnancy
* Active preoperative pulmonary infection
* Recent pulmonary infection (within 8 weeks)
* Active tobacco smoker
* Poorly controlled reactive airway disease (requires more than PRN albuterol)
* Non-Lung Protective Ventilation

Ages: 12 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients, both those that vape and those that do not, who meet the inclusion criteria and receive general anesthesia to facilitate surgical intervention at Naval Medical Center San Diego.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Perioperative pulmonary complications | From the initiation of general anesthesia through postoperative day seven.
  Complications of interest will include postoperative atelectasis with hypoxemia necessitating oxygen therapy, pneumothorax, pneumonia, bronchospasm, bronchospasm requiring bronchodilator therapy, exacerbation of underlying pulmonary disease, pneumonia, ARDS, and acute respiratory failure. Hospital course, including prolonged PACU stay, prolonged hospital admission for inpatients, and rate of ICU admissions, will also be investigated.

SECONDARY OUTCOMES:
Vaping cessation timeline | From the initiation of general anesthesia through postoperative day seven.
  Includes the relationship between vaping cessation timeline in the preoperative period and the occurrence of postoperative pulmonary complications

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No